CLINICAL TRIAL: NCT01728558
Title: Early Goal-Directed Sedation Compared With Standard Care in Mechanically Ventilated Critically Ill Patients: a Prospective Multicentre Randomised Controlled Trial
Brief Title: Early Goal-Directed Sedation Compared With Standard Care in Mechanically Ventilated Critically Ill Patients
Acronym: SPICE III RCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANZIC-RC/YS003
Record Dates: First submitted 2012-11-04; First posted 2012-11-20 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-04

CONDITIONS: Critical Illness and Mechanical Ventilation
Keywords: Sedation; Delirium; Goal Directed; Dexmedetomidine; Mortality; Mechanical ventilation; Intensive care; Critically Ill
MeSH Terms: conditions — Critical Illness; Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Goal Directed Sedation (Other): Early Goal Directed Sedation process of care involves:
  1. Early delivery of proposed intervention, shortly after initiating mechanical ventilation;
  2. Effective analgesia provided simultaneously and early (analgesia first).
  3. Regular and frequent assessment of patient wakefulness/sedative state;
  4. Avoidance of benzodiazepines and minimisation of use of propofol;
  5. Reduced overall sedation depth with targeted light sedation; Patients randomised to the EGDS arm will receive a sedative infusion of Dexmedetomidine withor without minimal propofol in order to maintain a RASS of -2 to +1.
  Dexmedetomidine infusion will be continued until sedation is no longer clinically indicated up to a maximum of 28 days after enrolment.
  Interventions: Other: Early goal Directed Sedation
- Standard care Sedation Arm (Active Comparator): Patients randomised to the standard care sedation arm will receive process of care sedation directed by the treating clinician. Based on the information from our observational study and the EGDS Pilot trial, most patients in this group are likely to receive midazolam and /or propofol. These agents will be infused to achieve the default target of Light sedation (RASS -2 to +1) whenever clinically appropriate and as specified by the treating clinician. The use remifentanil or dexmedetomidine for initial and maintenance sedation will be precluded.
  Interventions: Other: Standard care sedation

INTERVENTIONS:
Other: Early goal Directed Sedation
  Arms: Early Goal Directed Sedation
Other: Standard care sedation
  Arms: Standard care Sedation Arm

SUMMARY:
The Use of sedative drugs in intensive care is widespread. A cohort study conducted in Australia and New Zealand in 2010 revealed a high prevalence of deep sedation within the first 48 hours of mechanical ventilation which was independently linked to prolonged ventilation, hospital and 180 days mortality. Clinical practice is moving towards the use of lighter levels of sedation. Recent RCTs in Europe (JAMA 2012) and previous RCTs (JAMA 2009) supports growing evidence that dexmedetomidine facilitates rousable sedation, shortens ventilation time and attenuates delirium when compared to midazolam and propofol.

The investigators confirmed in a pilot study the feasibility, efficacy and safety of a process of care known as Early Goal Directed Sedation (EGDS) that delivers:

1. Early randomization after intubation or arrival in the ICU (intubated).
2. Early Adequate analgesia after randomization.
3. Goal directed sedation titrated to achieve light sedation.
4. Dexmedetomidine based algorithm as the primary sedative agent with avoidance of benzodiazepines.

The aim of this study is to assess the effectiveness of Early Goal Directed Sedation when compared to standard care sedation in critically ill patients.

The study hypothesis is that Early Goal-Directed Sedation (EGDS), compared to standard care sedation, reduces 90-day all-cause mortality in critically ill patients who require mechanical ventilation.

DETAILED DESCRIPTION:
This is a large-scale study into the effectiveness of a novel approach for sedation in ventilated critically ill patients. The primary aim of this study is to determine whether Early Goal Directed Sedation therapy, compared to standard care sedation, reduces 90-day mortality in critically ill patients ventilated > 24 hrs.

The study will be a randomized, unblinded, controlled trial conducted in approximately 35-50 intensive care units (ICUs) and will recruit 4000 mechanically ventilated patients (life support) who are expected to remain on the ventilator > 24 hours AND require immediate ongoing sedative medication for comfort, safety, and to facilitate the delivery of life support measures, including mechanical ventilation.

Patients with primary brain injury or prolonged weakness are excluded. Participants will be randomized into one of 2 study groups. All patients will receive adequate analgesia at randomization at the discretion of treating clinician. All randomized patients will have Light sedation as the default target unless otherwise clinically indicated. The intervention group will receive EGDS with dexmedetomidine as the primary sedative agent to achieve light sedation, with the addition of propofol as required. The use of benzodiazepines in the intervention group is not allowed, with the exception of specific, defined circumstances.

The control group will have sedation according to usual practice as chosen by the treating clinician. The use of dexmedetomidine is not allowed, with the exception of specific, defined circumstances.

Deidentified data will be collected and will include; Baseline demographic information; Doses of all sedative, analgesic and other related medications; Pain, sedation and delirium scores and major treatments such as ventilation time, tracheostomy and dialysis. Patients surviving to hospital discharge will be contacted by phone to determine independent survival status at 90 days and again at 180 days plus Health Related Quality of Life and cognitive function assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been intubated and is receiving mechanical ventilation
* The treating clinician expects that the patient will remain intubated until the day after tomorrow (unlikely to be extubated the following day).
* The patient requires immediate ongoing sedative medication for comfort, safety, and to facilitate the delivery of life support measures.

Exclusion Criteria:

* Age less than 18 years
* Patient is pregnant and/or lactating
* Has been intubated (excluding time spent intubated within an operating theatre or transport) for greater than 12 hours in an intensive care unit.
* Proven or suspected acute primary brain lesion such as traumatic brain injury, intracranial haemorrhage, stroke, or hypoxic brain injury.
* Proven or suspected spinal cord injury or other pathology that may result in permanent or prolonged weakness.
* Admission as a consequence of a suspected or proven drug overdose or burns.
* Administration of ongoing neuromuscular blockade.
* A mean arterial blood (MAP) pressure that is less than 50 mmHg despite adequate resuscitation and vasopressor therapy at time of randomisation
* Heart rate less than 55 beats per minute unless the patient is being treated with a beta-blocker or a high grade atrio-ventricular block in the absence of a functioning pacemaker.
* Known sensitivity to any of the study medications or the constituents of propofol (egg, soya or peanut protein)
* Acute fulminant hepatic failure
* Patient has been receiving full time residential nursing care.
* Death is deemed to be imminent or inevitable during this admission and either the attending physician, patient or substitute decision maker is not committed to active treatment.
* Patient has an underlying disease that makes survival to 90 days unlikely
* Patient has been previously enrolled in the SPICE study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Mortality | Day 90 post randomisation

SECONDARY OUTCOMES:
Ventilation free days | at 28 days following randomisation
Proportion of RASS measurements in target range | up to day 28
Incidence and duration of delirium measured by delirium free days | up to 28 days
Length of ICU stay | up to 180 days
Proportion of patients who receive a tracheostomy Proportion of patients who require: re-intubation, physical restraints,or unplanned extubation, | up to day 28
Cumulative dose of midazolam, propofol, dexmedetomidine, fentanyl, and morphine | up to 28 days
Duration of treatment with midazolam, propofol, dexmedetomidine, fentanyl, and morphine | up to 28 days
Mortality at hospital discharge | at hospital discharge up to 180 days
Length of hospital stay | up to 180 days
Readmission to ICU | at 90 days
EQ-5D questionnaire | at 180 days
Cognitive function | at 180 days
Mortality at ICU discharge | up to 180 days
Full time institutional dependency at 180 days | up to 180 days
Discharge destination | up to 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Yahya Shehabi, MD, FCICM, FANZCA, EMBA, Study Chair — University New South Wales, Prince of Wales Hospital, ANZIC-RC; Rinaldo Bellomo, Principal Investigator — ANZIC-RC & Austin Hospital; Steve A. R Webb, Principal Investigator — ANZIC-RC & Royal Perth Hospital; Michael C Reade, Principal Investigator — ANZIC-RC, Royal Brisbane & Women's Hospital, Department of Military Medicine and Surgery,; Belinda D Howe, Principal Investigator — ANZIC-RC; Ian M Seppelt, Principal Investigator — ANZIC-RC, Nepean Hospital; Colin McArthur, Principal Investigator — ANZIC-RC, Auckland Hospital; Simon Erikson, Principal Investigator — ANZIC-RC,; Lynne Murray, Principal Investigator — ANZIC-RC; Suhaini Kadiman, Principal Investigator — Institut Jantung Negara, Malaysia; Jukka Takala, Principal Investigator — Inselspital, Bern, Switzerland; Yaseen Arabi, Principal Investigator — King Abdulaziz Medical Centre, KSA; Matthew P Wise, Principal Investigator — University Hospital of Wales, UK
Locations (74):
- Australia (29):
  - Albury Hospital, Albury, New South Wales
  - Blacktown Hospital, Blacktown, New South Wales
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Hornsby Ku-ring-gai Hospital, Hornsby, New South Wales
  - Nepean Hospital, Penrith, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Darwin Hospital, Tiwi, Northern Territory
  - Sunshine Coast Hospital (Nambour Hospital), Buderim, Queensland
  - Royal Brisbane and Women's hospital, Herston, Queensland
  - Redcliffe Hospital, Redcliffe, Queensland
  - Gold Coast Hospital & Health Service, Southport, Queensland
  - Toowoomba Hospital, Toowoomba, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Lyell McEwan Hospital, Elizabeth Vale, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Launceston General Hospital, Launceston, Tasmania
  - Bendigo Hospital, Bendigo, Victoria
  - Dandenong Hospital, Dandenong, Victoria
  - Northern Hospital, Epping, Victoria
  - Geelong Hospital, Geelong, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
  - Central Gippsland Health Service, Sale, Victoria
  - Knox Private Hospital, Wantirna, Victoria
  - St John Of God, Subiaco, Perth, Western Australia
- Ireland (2):
  - St Vincent's University Hospital, Dublin, Dublin 4
  - St James's University Hospital, Dublin, Dublin 8
- Ospedale San Raffaele, Milan, Italy
- Malaysia (9):
  - Raja Perempuan Zainab II Hospital, Kota Bharu, Kelantan
  - Universiti Sains Malaysia Hospital, Kota Bharu, Kelantan
  - Penang General Hospital, George Town, Pulau Pinang
  - Queen Elizabeth Hospital, Kota Kinabalu, Sabah
  - Sarawak General Hospital, Kuching, Sarawak
  - Institut Jantung Negara, Kuala Lumpur
  - Kuala Lumpar General Hospital, Kuala Lumpur
  - University Malaya Medical Center, Kuala Lumpur
  - Melaka General Hospital, Malacca
- New Zealand (8):
  - Auckland City Hospital CVICU, Grafton, Auckland
  - Middlemore Hospital, Otahuhu, Auckland
  - Christchurch Hospital, Addington, Christchurch
  - North Shore Hospital, Takapuna, North Shore City
  - Wellington Hospital, Newtown, Wellington Region
  - Auckland City hospital, Auckland
  - Dunedin Hospital, Dunedin
  - Rotorua Hospital, Rotorua
- Saudi Arabia (3):
  - Prince Sultan Military Medical City, Riyadh
  - King Saud Medical City, Riyadh
  - King Abdulaziz Medical City, Riyadh
- Inselspital University Hospital Bern, Bern, Switzerland
- United Kingdom (21):
  - Kings College Hospital, Brixton, London
  - Freeman Hospital, High Heaton, Newcastle Upon Tyne
  - Queen Elizabeth Hospital King's Lynn, Kings Lynn, Norfolk
  - Derriford Hospital, Crownhill, Plymouth
  - University Hospital of North Tees, Hardwick, Stockton-on-Tees
  - Queen Elizabeth Hospital, Birmingham, Birmingham
  - Royal Bournemouth Hospital, Bournemouth
  - University Hospitals Bristol, Bristol
  - University Hospital of Wales, Cardiff
  - University Hospital of Coventry and Warwick, Coventry
  - Dorset County Hospital, Dorchester
  - Royal Infirmary of Edinburgh, Edinburgh
  - Western General Hospital, Edinburgh
  - Royal Liverpool University Hospital, Liverpool
  - St Thomas Hospital, London
  - St George's Hospital, London
  - University College Hospital, London
  - Altnagelvin Hospital, Londonderry
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Princess Royal University Hospital, Orpington
  - Royal Berkshire Hospital, Reading

REFERENCES:
- [Background] Shehabi Y, Bellomo R, Reade MC, Bailey M, Bass F, Howe B, McArthur C, Seppelt IM, Webb S, Weisbrodt L; Sedation Practice in Intensive Care Evaluation (SPICE) Study Investigators; ANZICS Clinical Trials Group. Early intensive care sedation predicts long-term mortality in ventilated critically ill patients. Am J Respir Crit Care Med. 2012 Oct 15;186(8):724-31. doi: 10.1164/rccm.201203-0522OC. Epub 2012 Aug 2. PMID 22859526
- [Derived] Shehabi Y, Serpa Neto A, Bellomo R, Howe BD, Arabi YM, Bailey M, Bass FE, Bin Kadiman S, McArthur CJ, Reade MC, Seppelt IM, Takala J, Wise MP, Webb SA; SPICE III Study Investigators. Dexmedetomidine and Propofol Sedation in Critically Ill Patients and Dose-associated 90-Day Mortality: A Secondary Cohort Analysis of a Randomized Controlled Trial (SPICE III). Am J Respir Crit Care Med. 2023 Apr 1;207(7):876-886. doi: 10.1164/rccm.202206-1208OC. PMID 36215171
- [Derived] Cioccari L, Luethi N, Bailey M, Shehabi Y, Howe B, Messmer AS, Proimos HK, Peck L, Young H, Eastwood GM, Merz TM, Takala J, Jakob SM, Bellomo R; ANZICS Clinical Trials Group and the SPICE III Investigators. The effect of dexmedetomidine on vasopressor requirements in patients with septic shock: a subgroup analysis of the Sedation Practice in Intensive Care Evaluation [SPICE III] Trial. Crit Care. 2020 Jul 16;24(1):441. doi: 10.1186/s13054-020-03115-x. PMID 32678054
- [Derived] Shehabi Y, Howe BD, Bellomo R, Arabi YM, Bailey M, Bass FE, Bin Kadiman S, McArthur CJ, Murray L, Reade MC, Seppelt IM, Takala J, Wise MP, Webb SA; ANZICS Clinical Trials Group and the SPICE III Investigators. Early Sedation with Dexmedetomidine in Critically Ill Patients. N Engl J Med. 2019 Jun 27;380(26):2506-2517. doi: 10.1056/NEJMoa1904710. Epub 2019 May 19. PMID 31112380
- [Derived] Moore JPR, Anstey C, Murray L, Fraser JF, Singer M. Allostasis and sedation practices in intensive care evaluation: an observational pilot study. Intensive Care Med Exp. 2018 Jun 20;6(1):13. doi: 10.1186/s40635-018-0179-0. PMID 29926288